CLINICAL TRIAL: NCT03672578
Title: Reducing Sugar-sweetened Beverage Consumption Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1124060; 1K01DK113068-01A1 (NIH)
Record Dates: First submitted 2018-09-10; First posted 2018-09-14 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Intention; Health Knowledge, Attitudes, Practice
Keywords: Diet; Young Adults; Health messaging
MeSH Terms: conditions — Behavior | interventions — icon infiltrant

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Loss-frame, text-only, no attribution (Experimental): Label participants will see is loss-frame, text-only, and with no attribution
  Interventions: Other: loss-frame; Other: text-only; Other: no attribution
- Gain-frame, text-only, no attribution (Experimental): Label participants will see is gain-frame, text-only, and with no attribution
  Interventions: Other: gain-frame; Other: text-only; Other: no attribution
- Loss-frame, icon, no attribution (Experimental): Label participants will see is loss-frame, icon, and with no attribution
  Interventions: Other: loss-frame; Other: icon; Other: no attribution
- Grain-frame, icon, no attribution (Experimental): Label participants will see is gain-frame, with an icon, and with no attribution
  Interventions: Other: gain-frame; Other: icon; Other: no attribution
- Loss-frame, icon, attribution (Experimental): Label participants will see is loss-frame, icon, and with attribution
  Interventions: Other: loss-frame; Other: icon; Other: attribution
- Gain-frame, icon, attribution (Experimental): Label participants will see is grain-frame, icon, and with attribution
  Interventions: Other: gain-frame; Other: icon; Other: attribution
- Loss-frame, text-only, attribution (Experimental): Label participants will see is loss-frame, text-only, and with attribution
  Interventions: Other: loss-frame; Other: text-only; Other: attribution
- Gain-frame, text-only, attribution (Experimental): Label participants will see is gain-frame, text-only, and with attribution
  Interventions: Other: gain-frame; Other: text-only; Other: attribution
- No label (Placebo Comparator): Participant will not see a label
  Interventions: Other: No label

INTERVENTIONS:
Other: loss-frame — loss frame label
  Arms: Loss-frame, icon, attribution; Loss-frame, icon, no attribution; Loss-frame, text-only, attribution; Loss-frame, text-only, no attribution
Other: gain-frame — gain frame label
  Arms: Gain-frame, icon, attribution; Gain-frame, text-only, attribution; Gain-frame, text-only, no attribution; Grain-frame, icon, no attribution
Other: text-only — text-only label
  Arms: Gain-frame, text-only, attribution; Gain-frame, text-only, no attribution; Loss-frame, text-only, attribution; Loss-frame, text-only, no attribution
Other: icon — label with icon and text
  Arms: Gain-frame, icon, attribution; Grain-frame, icon, no attribution; Loss-frame, icon, attribution; Loss-frame, icon, no attribution
Other: attribution — label with attribution
  Arms: Gain-frame, icon, attribution; Gain-frame, text-only, attribution; Loss-frame, icon, attribution; Loss-frame, text-only, attribution
Other: no attribution — label with no attribution
  Arms: Gain-frame, text-only, no attribution; Grain-frame, icon, no attribution; Loss-frame, icon, no attribution; Loss-frame, text-only, no attribution
Other: No label — No label
  Arms: No label

SUMMARY:
This study aims to test sugar-sweetened beverage (SSB) health labeling elements in an online experiment to determine which elements are the most salient among young adults.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years of age
* current/recent (<1 year of graduation) undergraduate student at 3 specific universities
* English-speaking
* consumes at least 2 SSBs per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2971 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-11-17 (Actual)

PRIMARY OUTCOMES:
SSB Intention | Up to 20 minutes
  Intention to consume SSBs measured by hypothetical selection of a beverage from images of beverage options.

SECONDARY OUTCOMES:
SSB Intention (2) | Up to 20 minutes
  Measured by survey items assessing intention to consume SSBs on a scale from 1 (not at all likely) to 7 (extremely likely).
SSB attitudes | Up to 20 minutes
  Measured by survey items assessing perceived healthfulness of SSBs on a scale from 1 (extremely unhealthy) to 7 (extremely healthy).
SSB knowledge | Up to 20 minutes
  Measured by survey items assessing knowledge of number of calories (estimate provided by participant) and sugar (estimated by participant, in teaspoons) contained in SSBs.
SSB norms | Up to 20 minutes
  Measured by survey item assessing how often participants perceive their peers to consume SSBs (1 = multiple times a day, 2 = daily, 3 = weekly, 4 = less than once a week, and 5 = never) and item on perception that people who are important to the participant would want them to limit SSB intake, on a scale from 1 (not at all) to 5 (completely) .

OTHER OUTCOMES:
SSB self-efficacy | Up to 20 minutes
  Measured by survey item assessing how confident participant feels in reducing SSB consumption, on a scale from 1 (not at all) to 5 (completely).
Social interaction | Up to 20 minutes
  Measured by survey item assessing likelihood participant will encourage others to reduce SSB consumption, on a scale from 1 (not at all) to 5 (completely).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, ScD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No